CLINICAL TRIAL: NCT04725487
Title: Community With Immigrants - a Step on the Road to Employment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Absalon (Other)
Collaborators: Naestved Municipality (Unknown); Danish Refugee Council (Unknown); Den A.P. Møllerske Støttefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCAbsalon
Record Dates: First submitted 2020-12-18; First posted 2021-01-26 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2021-01

CONDITIONS: Health Knowledge; Attitude to Health; Practice
Keywords: Refugee families; Social and health promoting intervention; Well-being; Employment; Integration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard integration program with social and health promoting intervention (Experimental): Participants follow the standard integration program offered by Naestved Municipality and participate in various social and health promoting activities in addition
  Interventions: Other: Standard integration program with social and health promoting intervention
- Standard integration program (Active Comparator): Participants follow the standard integration program offered by Naestved Municipality
  Interventions: Other: Standard integration program

INTERVENTIONS:
Other: Standard integration program with social and health promoting intervention — * Basic language course, internships, courses in Labour market knowledge and Danish culture
  * Physical activity workshops
  * Community gardening (garden workshops)
  * Entrepreneurship course
  * MindSpring course
  * Family excursions
  * Danish language workshops
  Arms: Standard integration program with social and health promoting intervention
Other: Standard integration program — Standard integration program (basic language course, internships, courses in Labour market knowledge and Danish culture)
  Arms: Standard integration program

SUMMARY:
The study will investigate if a standard integration programme in combination with a social and health promoting intervention can increase health and well-being among refugee families and influence success with education and employment.

DETAILED DESCRIPTION:
Increased health and well-being can lead to stronger motivation and ability to get involved in education or employment and thereby improve integration of refugee families.

The aim of the study is to investigate the effect of various social and health promoting activities such as physical activity workshops, community gardening, entrepreneurship training, MindSpring course, family excursions and language education on health, well-being, social relations and success with job and education. Increased success with self-sufficiency can support action competence and play a key role in the integration process. Outcome measures are based on self-reporting, biological measures and municipal registry data.

ELIGIBILITY:
Inclusion Criteria:

* Adult refugees aged 18 years and above
* Young refugees aged 13 -17 years
* Must have obtained Danish asylum and live in Naestved Municipality

Exclusion Criteria:

* Physical and/or mental illness which prevents the individual from participating in the integration program offered by Naestved Municipality
* Illness which does not allow collection of a venous blood sample and saliva sample.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The Warwick-Edinburgh Mental Well-Being Scale - 7 items (WEMWBS) | Change from baseline to 12 months and 24 months
  WEMWBS is a validated measure of mental well-being and contains seven questions (a shortened version of the WEMWBS - 14 items). The scoring range for each item is from 1- 5, and the total score is from 7-35. The seven items have superior scaling properties to the 14 items, and mean raw scores are therefore transformed to metric scores using a standard conversion table.
Mean change from baseline in self-reported health | Change from baseline to 12 months and 24 months
  General health is assessed based on a question on self-reported health in the SF-12 questionnaire (a 12-Item short form health survey). SF 12 is a short version of the generic questionnaire SF 36 that measures health-related quality of life in the past four weeks.
  Scoring range is between 1-5 points. Mean score is calculated at baseline, 12 months and 24 months.
Mean change from baseline in cortisol, nmol/L | Change from baseline to 24 months
  Cortisol measured in saliva
Mean change from baseline in blood sugar (HBA1C), mmol/mol | Change from baseline to 24 months
  Blood sugar measured in venous blood
Mean change from baseline in total cholesterol, mmol/L | Change from baseline to 24 months
  Total cholesterol measured in venous blood
Mean change from baseline in self-reported social relations | Change from baseline to 12 months and 24 months
  Social relations are assessed based on five questions from the National Health Profile Survey (used in the Danish National Health Survey) in combination with one self-formulated question regarding contact with family members, friends, colleagues, neighbors and friends from social medias. Scoring range is between 1-5 points. Mean score is calculated at baseline, 12 months and 24 months.
Change in employment status | Change from baseline to 12 months and 24 months
  From unemployed to employed; from not being involved in education to being involved in education. Data from municipal registers.

SECONDARY OUTCOMES:
Mean change from baseline in Dihydepiandrosteron-sulfate (DHEAS), µmol/L | Change from baseline to 24 months
  DHEAS measured in venous blood
Mean change from baseline in interleukin-6 (IL-6), ng/L | Change from baseline to 24 months
  IL-6 measured in venous blood
Mean change from baseline in C-reactive protein (CRP), nmol/L | Change from baseline to 24 months
  CRP measured in venous blood
Mean change from baseline in fibrinogen (FIBR), g/L | Change from baseline to 24 months
  FIBR measured in venous blood
Mean change from baseline in weight | Change from baseline to 24 months
  Weight (in kilograms). Weight is measured in kilograms
Mean change from baseline in BMI | Change from baseline to 24 months
  Weight and height (measured in meters) will be combined to report BMI in kg/meters2
Mean change from baseline in blood pressure | Change from baseline to 24 months
  Systolic and diastolic blood pressure (mmHg) will be measured using the Omron M3 blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Nina O Nielsen, Ph.d, Principal Investigator — University College Absalon (UCAbsalon)
Locations (1):
- Nina Odgaard Nielsen, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No